CLINICAL TRIAL: NCT05333445
Title: Assessing the Nurse-led Educational Intervention in Patients Undergoing Catheter Ablation for Atrial Fibrillation: a Randomized Controlled Trial
Brief Title: NURSE-led Follow-up in Patients Undergoing CATheter Ablation for Atrial Fibrillation
Acronym: NURSECAT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Head of Arrythmia Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURSECAT-AF
Record Dates: First submitted 2022-03-25; First posted 2022-04-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; nurse-led; educational intervention; risk factors; quality of life
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nursing intervention (Experimental): The NI will be performed at 3 times: face to face between 21 and 7 days before admission, between 7 and 15 days after the date of ablation, and 6 months after the ablation procedure.
  Interventions: Behavioral: educational program; Behavioral: risk factors management; Behavioral: telephone and e-mail contact
- control group (Active Comparator): After hospital discharge, all patients will be referred to their primary care physician or cardiologist for follow-up.
  Patients will receive standard follow-up checks by the medical team will not receive structured education from the nurse.
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: educational program — Education for the management of AF is carried out in a structured way, following the Bowyer model using the following pre-specified subtitles: "How the heart works"; "Causes and risk factors of AF"; "Symptoms of AF";"" Goals of treatment in atrial fibrillation ""; ''preparation for the ablation procedure''; and "Lifestyle Modification". The technique consists of discussing the main subtitles and adapting the visit line to the needs of each patient
  Arms: Nursing intervention
Behavioral: risk factors management — identify risk factors and offer guidance based on management strategies for the specific risk factor in each case
  Arms: Nursing intervention
Behavioral: telephone and e-mail contact — patients will also be provided with a phone number and email to contact the nurse for any concerns outside the designated times within the twelve-month follow-up.
  Arms: Nursing intervention
Other: usual care — standard care
  Arms: control group

SUMMARY:
The study aims to examine the effect of nurse-led education program on quality of life, atrial fibrillation (AF) risk factors, AF symptomatology, arrhythmia recurrence rate, and readmission rate after AF catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* Derivatives from the outpatient clinic of the center itself, as well as patients referred from other centers that have ours as a reference for a first AF ablation procedure.
* Have signed the informed consent.

Exclusion Criteria:

* Patients with cognitive impairment or disorientation.
* Patients with problems of comprehension or expression of Spanish or Catalan.
* Patients who are part of the medical or nursing group.
* Patient with defined heart failure with a left ventricular ejection fraction (LVEF) less than 40% and a NYHA III or IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
changes from the baseline and better score in the validated ASTA questionnaire of the intervention group compared to the control group at 12 months in quality of life of patients . | 12 months
  We will use the second part of ASTA questionnaire: it consists of 13 questions and the answers are measured using a Likert frequency scale from "Never = 0" to "Always = 4". Higher scores on this scale represent poorer quality of life.

SECONDARY OUTCOMES:
number of patients who have the AF risk factor within normal parameters | 12 months
  differences between the two groups in number of patients with BMI and/or waist circumference changes from the baseline, better score on the Minnesota Adapted Scale for Physical Exercise, number of patients who do not smoke or drink alcohol, number of patients with positive polysomnography, number of patients with impaired of the analytical parameters of HbA1c, TSH, LDL or Triglycerides.
number of participants with re-hospitalisation or emergency room visits for cardiovascular cause | 12 months
  differences between the two groups in number of patients who come to the emergency room or re-admit after discharge from catheter ablation.
number of participants with recurrences at AF rhythm | 12 months
  number of AF detected by ECG or 24-hour cardiac holter routine at 3, 6 and 12 months.
differences between both groups in the score received by the patients in the User Experience Questionnaire based on the Picker-33 Patient Experience Questionnaire | 3 months
  It consists of 14 closed-ended questions and is performed using a checklist to assign numerical values to subjective satisfaction using a Likert scale from "No = 0" to "Yes, always = 4". Higher scores on this scale represent greater satisfaction. An open question has been added so that participants can add their suggestions
Differences between both groups in intensity, frequency and severity of symptoms related to AF evaluated with the validated ASTA questionnaire | 12 months
  differences between both groups in the score obtained in the first part of the validated questionnaire in Spanish and English sensitive for patients with AF. It will be self-filled by the patient himself. It consists of 8 questions formulated in 3 different ways: (1) Multiple correct answer multiple choice questions. (2) Multiple choice questions with only one correct answer. (3) Checklist for assigning numerical values to frequency using a Likert scale from "Never = 0" to "Always = 4". Higher scores on this scale represent greater severity of symptoms.
differences between both groups in the score obtained in the adapted AFKAT questionnaire patient's knowledge of AF. | 3 months
  differences between both groups in the Level of knowledge of FA through the AFKAT questionnaire validated in English but adapted and translated into Spanish by our team. It consists of 25 questions with dichotomous True/False answers. The more true answers, the better knowledge the participant has.
calls and emails received | 12 months
  Quantify the calls and emails received from patients to the FA nurse.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, barcelona, Spain